CLINICAL TRIAL: NCT05324319
Title: Single Blinded Randomized Controlled Trial on BNT162b2 or mRNA-1273 (mRNA) vs Ad26COVS1 or ChAdOx1-S (Viral Vector) for Third Vaccination in Kidney Transplant Recipients Without SARS-CoV-2 Spike Protein Antibodies Following Full Vaccination
Brief Title: Homologous vs Heterologous Third Vaccination in Kidney Transplant Recipients Kidney Transplant Recipients
Acronym: BOOST_TX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Roman Reindl-Schwaighofe, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BOOST_TX
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ad26COVS1; BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- homologous 3rd vaccination (mRNA vaccine) (Active Comparator): Participants will receive a third SARS-CoV-2 vaccination with the same mRNA vaccine they received for the initial prime-boost vaccination (BNT162b2 or mRNA-1273 )
  Interventions: Drug: BNT162B2; Drug: mRNA-1273
- heterologous 3rd vaccination (vector vaccine) (Experimental): participants will receive a third SARS-CoV-2 vaccination with a vector vaccine (Ad26COVS1 or ChAdOx1-S)
  Interventions: Drug: Ad26COVS1; Drug: ChAdOx1 SARS2 Vaccine

INTERVENTIONS:
Drug: Ad26COVS1 — Heterologous vaccination
  Arms: heterologous 3rd vaccination (vector vaccine)
Drug: ChAdOx1 SARS2 Vaccine — Heterologous vaccination
  Arms: heterologous 3rd vaccination (vector vaccine)
Drug: BNT162B2 — Homologous vaccination
  Arms: homologous 3rd vaccination (mRNA vaccine)
Drug: mRNA-1273 — Homologous vaccination
  Arms: homologous 3rd vaccination (mRNA vaccine)

SUMMARY:
Randomized-controlled trial comparing homologous (mRNA vaccine) vs. heterologous (vector vaccine) for third SARS-CoV-2 vaccine dose in kidney transplant recipients not responding to initial prime-boost vaccination with an mRNA vaccine.

ELIGIBILITY:
Inclusion Criteria:

* patient has received a kidney transplantation
* full SARS-CoV-2 vaccination with mRNA vaccine (two doses) at least 4 weeks before screening
* > 18 years of age
* no SARS-CoV-2 spike protein antibodies at least 4 weeks after the second dose of an mRNA vaccine

Exclusion Criteria:

* acute illness with fever
* Prior documented infection with SARS-CoV-2
* triple anticoagulation therapy
* Subject is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s)
* Subject has known sensitivity or intolerance to any of the products to be administered for the purpose of this study
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with the study procedures
* Subject is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Seroconversion at 4 weeks | 4 weeks
  number of patients developing SARS-CoV-2 antibodies at 4 weeks after 3rd vaccination

SECONDARY OUTCOMES:
Seroconversion at 12 weeks | 3 months
  number of patients developing SARS-CoV-2 antibodies at 12 weeks after 3rd vaccination (> 0.8 BAU/mL)
SARS-CoV-2 antibody levels at 4 weeks | 4 weeks
  SARS-CoV-2 antibody levels at 4 weeks after the third vaccination
SARS-CoV-2 antibody levels at 12 weeks | 3 months
  SARS-CoV-2 antibody levels at 12 weeks after the third vaccination
Seroconversion at 36 weeks | 6 months
  number of patients developing SARS-CoV-2 antibodies at 36 weeks after 3rd vaccination (> 0.8 BAU/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Medicial University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided